CLINICAL TRIAL: NCT05152420
Title: A Randomised, Double-Blind, Placebo-Controlled, Single Ascending Dose Trial to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenously Administered VMX-C001 in Healthy Subjects (Part 1) and in Combination With Selected Direct Oral Anticoagulants (DOACs) in Healthy Older Subjects (Part 2)
Brief Title: Study of Intravenous VMX-C001 in Healthy Subjects and in Combination With Selected Direct Oral Anticoagulants in Healthy Older Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VarmX B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMX-C001-01
Record Dates: First submitted 2021-11-17; First posted 2021-12-09 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Coagulation Disorder
Keywords: Direct oral anticoagulant (DOAC); Human coagulation factor X
MeSH Terms: conditions — Hemostatic Disorders | interventions — apixaban; Rivaroxaban; edoxaban

STUDY DESIGN:
Intervention Model Description: Placebo controlled, single ascending dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1 - Cohort 1 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 1 - Cohort 2 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 1 - Cohort 3 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 1 - Cohort 4 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 1 - Cohort 5 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 1 - Cohort 6 (Experimental): Single dose cohort
  Interventions: Drug: VMX-C001; Drug: Placebo
- Part 2 - Cohort 1 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 2 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 3 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 4 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 5 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 6 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Part 2 - Cohort 7 (Experimental): Single dose cohort of selected FXa DOAC anticoagulant in combination with VMX-C001
  Interventions: Drug: VMX-C001; Drug: Placebo; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban

INTERVENTIONS:
Drug: VMX-C001 — VMX-C001 is human factor X engineered to be insensitive to factor Xa DOACs
Drug: Placebo — VMX-C001 matched placebo
Drug: Apixaban — FXa Inhibitor
  Arms: Part 2 - Cohort 1; Part 2 - Cohort 2; Part 2 - Cohort 3; Part 2 - Cohort 4; Part 2 - Cohort 5; Part 2 - Cohort 6; Part 2 - Cohort 7
Drug: Rivaroxaban — FXa Inhibitor
  Arms: Part 2 - Cohort 1; Part 2 - Cohort 2; Part 2 - Cohort 3; Part 2 - Cohort 4; Part 2 - Cohort 5; Part 2 - Cohort 6; Part 2 - Cohort 7
Drug: Edoxaban — FXa Inhibitor
  Arms: Part 2 - Cohort 1; Part 2 - Cohort 2; Part 2 - Cohort 3; Part 2 - Cohort 4; Part 2 - Cohort 5; Part 2 - Cohort 6; Part 2 - Cohort 7

SUMMARY:
A single centre, double-blind, randomized, parallel group, placebo-controlled study in healthy subjects conducted in two parts:

Part 1: Single ascending doses in healthy subjects aged 18 to 49 years to assess safety, pharmacokinetics (PK) and pharmacodynamic (PD) effects of VMX-C001.

Part 2: Healthy subjects aged 50 to 79 years to assess safety, PK and PD effects of VMX-C001 in the presence of DOACs.

ELIGIBILITY:
Inclusion Criteria:

1. In Part 1, men and women of any ethnic origin aged between 18 and 49 years of age, inclusive, at the time of Screening.
2. In Part 2, men and women of any ethnic origin aged between 50 and 79 years of age, inclusive, at the time of Screening.
3. Male subjects must be willing to use appropriate contraception, such as a condom, and to refrain from sperm donation during the study and until 90 days after study drug administration.
4. Women of child-bearing potential must agree not to attempt to become pregnant and to use a highly effective form of birth control during the study and for 90 days after study drug administration when their sexual partner has not been vasectomized. Highly effective forms of birth control entail the use of combined (estrogen- and progestogen-containing) or progestogen-only hormonal contraception associated with inhibition of ovulation, an intrauterine device (IUD), an intrauterine hormone-releasing system (IUS) or abstinence.
5. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with documented follicle-stimulating hormone (FSH) ≥30 milli-International units (mIU)/mL).
6. Surgically sterile women are defined as those who have had a surgical bilateral oophorectomy with or without hysterectomy, total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, the reproductive status of the woman has to be confirmed by follow-up hormone level assessment. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
7. All women must have a negative pregnancy test result at Screening and on Day -1.
8. Subject must weigh between 60 and 120 kg, inclusive, and must have a BMI between 18.0 and 30.0 kg/m^2, inclusive, at Screening and on Day -1.
9. Subject must be in good health, as determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations (congenital non hemolytic hyperbilirubinemia is acceptable).
10. Participant is willing and able to give their written informed consent to participate in the study and to abide by the study restrictions.
11. Participant has good upper limb venous access.

Exclusion Criteria:

1. The participant has taken piroxicam in the two weeks prior to the first administration of study drug or DOAC.
2. The participant has taken any non-aspirin non-piroxicam NSAID in the week prior to the first administration of study drug or DOAC.
3. The participant requires or has taken during the month prior to first administration of study drug or DOAC, vitamin K for therapeutic reasons. Vitamin K not taken for therapeutic purposes is acceptable, e.g. as part of a multivitamin supplement.
4. The participant is receiving or requires, for any cause, any anticoagulant or antiplatelet therapy including warfarin, clopidogrel or aspirin or any other anticoagulant or antiplatelet agent or has used these therapies in the month prior to the first administration of study drug or DOAC.
5. The participant has received any prescribed oral, systemic or topical medication, including coronavirus disease (COVID)-19 vaccination, within 14 days prior to the first administration of study drug or DOAC (with the exception of contraceptives), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
6. The participant has used any non-prescribed systemic or topical medication (including herbal remedies) within one week prior to the first administration of study drug or DOAC (with the exception of oral vitamin/mineral supplements (that do not contain vitamin k) and paracetamol), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
7. The participant is currently participating in a clinical study, e.g. attending follow-up visits or has been administered an investigational drug (new chemical or biological entity) in the 3 months prior to administration of the study drug.
8. The participant has donated >500 mL blood, plasma or platelets in the 3 months prior to Screening.
9. Because of an increased risk of thrombosis participants with known diabetes mellitus or a fasted glucose ≥7.0 mmol/l at Screening.
10. The participant has any bleeding diathesis, any increased risk of bleeding or, in the opinion of the Principal Investigator, is at increased risk of the consequences of bleeding including but not limited to the following:

    1. gastro-intestinal ulceration within the last 3 months
    2. known or suspected oesophageal varices.
    3. vascular aneurysms or known arteriovenous malformations;
    4. history of known major intraspinal or intracerebral vascular abnormalities.
    5. history of brain, spinal or ophthalmic surgery within the last year.
    6. any intracranial hemorrhage.
    7. uncontrolled severe hypertension.
11. The participant has, in the opinion of the Principal Investigator, any increased risk of thrombosis or thromboembolism including any known thrombophilia, such as antiphospholipid syndrome, or any past history of thrombosis.
12. The participant has a significant history of drug allergy, as determined by the Principal Investigator.
13. The participant has, at Screening or on Day -1, a supine blood pressure or supine pulse rate ≥ 150/95 mmHg and 100 beats per minute (bpm), respectively, or < 90/40 mmHg and 40 bpm, respectively, confirmed by a repeat assessment.
14. The participant consumes >21 alcoholic drinks/week for men or >14 alcoholic drinks/week for women (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1 measure [25 mL] of spirits), or has a significant history of alcoholism or drug/chemical abuse, as determined by the Principal Investigator for Part 1. For Part 2, the participant consumes >7 alcoholic drinks/week.
15. The participant has a positive urine drug screen, alcohol breath test or cotinine test results at Screening or on Day -1, confirmed by repeat testing.
16. The female participant has a positive pregnancy test at Screening or on Day -1 or is lactating.
17. The participant currently smokes or uses nicotine-containing products. Former smokers will be eligible, provided participants have not smoked for at least 3 months prior to administration of the study drug.
18. The participant has, or has a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological or other major disorders, as determined by the Principal Investigator.
19. The participant has a positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody test result at Screening.
20. The participant has an abnormality in the 12-lead ECG at Screening or on Day -1 that, in the judgement of the Principal Investigator may, during the study, interfere with the interpretation of 12-lead ECG results, including average QTcF interval >450 msec for men or >470 msec for women, 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as average PR<110 msec, confirmed by a triplicate repeat ECG.
21. The participant has any other condition that, in the opinion of the Principal Investigator, would compromise the safety of the participant or the participant's ability to comply with the protocol and complete the study.
22. The participant has renal insufficiency (serum creatinine level > 1.25 times upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) of ≤60 mL/minute).
23. The participant has active liver disease (ALT/ aspartate aminotransferase (AST) >1.5x ULN, total bilirubin > 1.5x ULN at Screening or on Day -1. One re-test is allowed).

    Additional exclusion criteria for Part 2 only:
24. Because of an effect on DOACs,participants are to be excluded if he/she receives or has received medication that is an inhibitor of P-glycoprotein or CYP3A4. (eg clarithromycin, erythromycin and azole-antimycotics such as ketoconazole, itraconazole, voriconazole and osaconazole or HIV protease inhibitors.) within 30 days prior to first administration of DOAC.
25. Because of an effect on DOACs, participants are to be excluded if he/she receives or has received treatment with CYP3A4 inducers (eg St. John's wort, rifampicin, phenytoin, carbamazepine, phenobarbital within 30 days prior to first administration of DOAC.
26. Because of an effect on DOACs, participants are to be excluded if he/she receives or has received treatment with selective serotonin reuptake inhibitors (SSRIs) or selective noradrenaline reuptake inhibitors (SNRIs) within 30 days prior to first administration of DOAC.
27. The participant has any contra-indication to treatment with DOACs.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part 1) | Up to Day 28
  Number of Subjects with One or More Drug Related Adverse Events (AEs) or any Serious AEs
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part 2) | Up to Day 31
  Number of Subjects with One or More Drug Related Adverse Events (AEs) or any Serious AEs
PK of VMX-C001 in plasma after single dose administration - Cmax (Part 1) | Up to Day 7
  Maximal concentration
PK of VMX-C001 in plasma after single dose administration - tmax (Part 1) | Up to Day 7
  Time of maximal concentration
PK of VMX-C001 in plasma after single dose administration - t1/2 (Part 1) | Up to Day 7
  Terminal elimination half-life
PK of VMX-C001 in plasma after single dose administration - AUC0-last (Part 1) | Up to Day 7
  Area under the concentration-time curve from time of dosing to last measurable concentration
PK of VMX-C001 in plasma after single dose administration - AUC0-inf (Part 1) | Up to Day 7
  Area under the concentration-time curve from time of dosing extrapolated to infinity
PK of VMX-C001 in plasma after single dose administration - Lambda z (Part 1) | Up to Day 7
  Terminal elimination rate constant
PK of VMX-C001 in plasma after single dose administration - CL (Part 1) | Up to Day 7
  Total body clearance
PK of VMX-C001 in plasma after single dose administration - Dose proportionality (Part 1) | Up to Day 7
Change in D-dimer, Thrombin-Antithrrombin complexes and prothrombin fragments F1 and F2 following dosing with VMX-C001 (Part 1 and Part 2) | Up to Day 28 post dose with VMX-C001
Change from baseline in thrombin generation (ETP) following dosing with VMX-C001 in subjects previously dosed with DOAC anticoagulants (Part 2) | Up to 24 hours post dose with VMX-C001
DOAC plasma concentrations (Part 2) | Up to Day 5

SECONDARY OUTCOMES:
Antibodies against VMX-C001 in plasma (Part 1) | Up to Day 28
  Immunogenicity
Antibodies against VMX-C001 in plasma (Part 2) | Up to Day 31
  Immunogenicity
Antibodies against human coagulation FX in plasma (Part 1) | Up to Day 28
  Immunogenicity
Antibodies against human coagulation FX in plasma (Part 2) | Up to Day 31
  Immunogenicity

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No